CLINICAL TRIAL: NCT05326477
Title: Predictors of Behavioral Obesity Treatment Outcomes
Acronym: REBOOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20042007
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard-of-care behavioral weight loss treatment (Other): 6-months of group-based behavioral weight loss treatment following the Centers for Disease Control and Prevention Prevent T2 curriculum.
  Interventions: Behavioral: Behavioral weight loss treatment

INTERVENTIONS:
Behavioral: Behavioral weight loss treatment — The weight loss intervention consists of the first 6 months of the Centers for Disease Control and Prevention's Prevent T2 program.

SUMMARY:
Socioceconomically disadvantaged individuals typically have poor outcomes in behavioral weight loss interventions, but the reasons for this are unknown. This project will characterize the mechanisms through which adverse daily experiences and present bias -- a cognitive adaptation to harsh and unpredictable environments -- account for disparities in weight loss outcomes.

DETAILED DESCRIPTION:
Individuals of lower socioeconomic status (SES) lose only half as much weight in behavioral weight loss interventions as those of higher SES. This is a clinically meaningful difference in outcomes that has been consistently documented. The overarching aim of this project is to identify the mechanisms that account for SES-related disparities in behavioral weight loss outcomes, which would enable the development of more effective obesity treatment approaches for lower SES populations. One potential mechanism is present bias, which is a tendency to focus on one's immediate needs that may result from exposure to harsh and unpredictable environments. Present bias is a compelling candidate as a mechanism of SES-related disparities in weight loss outcomes because it is much more pronounced in lower SES populations, and it has been linked to obesity risk, maladaptive eating behaviors, and poor diet quality. A second set of potential mechanisms includes adverse daily experiences such as stress, cognitive demands, and exposure to tempting foods. Stress and cognitive demands are more prevalent or severe in the lives of lower SES populations, and can disrupt the executive functions that are important for adhering to weight control behaviors during obesity treatment.

This project will allocate equal numbers of subjects of lower and higher SES to a standard-of-care weight loss intervention. Importantly, the SES groups will be balanced with respect to ethnic/racial minority status. Weight loss outcomes and adherence to three key weight control behaviors (dietary lapses, dietary self-monitoring, and physical activity) will be rigorously measured across six months of follow up. Individual differences in present bias will be thoroughly assessed at baseline. Ecological momentary assessment will be used to capture exposure to adverse daily experiences, as well as momentary changes in present bias. Aim 1 is to test whether present bias accounts for SES-related disparities in behavioral weight loss outcomes and adherence to key weight control behaviors. Aims 2a and 2b will characterize the role of adverse daily experiences in SES-related disparities in weight loss outcomes and adherence to weight control behaviors, both overall and among present-biased individuals in particular. Aim 3 is to explore the contribution of race to SES-related disparities in weight loss outcomes, which has been challenging to elucidate in prior studies due to significant confounding of race and SES at the societal level. The results of this study could lead to a new understanding of how socioeconomic disadvantage impacts adherence to behavioral treatment for obesity, and suggest entirely new treatment approaches focused on mitigating present bias or delivering tailored intervention content during "moments of risk" for lapses in adherence.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Obesity (body mass index ≥30 kg/m2)
3. Meets criteria for either the lower SES or higher SES cohort

Exclusion Criteria:

1. Not fluent in English
2. Change in income or financial assets exceeding ±75% of federal poverty guideline within the past 12 months, or expected in the next 6 months, if this change would result in reclassification on SES.
3. Previous or planned bariatric surgery, or concurrent engagement in other behavioral or pharmacological treatment for obesity
4. Resides more than 20 miles away from Rush, or planning to move outside of this geographic area during the study period
5. Body mass index ≥60 kg/m2, due to increased injury risk with exercise
6. History of bariatric surgery, or current engagement in another weight loss therapy
7. Lack of reliable access to cell or landline phone
8. Medical contraindications to treatment, including osteoporosis, cognitive impairment (Montreal Cognitive Assessment ≤25), active substance abuse based on the World Health Organization's ASSIST screener, lack of physician clearance for participation, or serious medical illness (e.g., stage 3 or 4 heart failure, cancer, renal failure, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Weight change | Months 2, 4, and 6
  Weight change, reported as a percentage of baseline weight

SECONDARY OUTCOMES:
Adherence to dietary self-monitoring | Months 2, 4, and 6
  Adherence to daily dietary self-monitoring will be scored as a binary variable (adherent vs. non-adherent) based on whether a subject recorded ≥50% of prescribed daily calorie intake goal on a given day. For example, an individual with a goal of 1350 kcal/d would be considered adherent on days in which at least 675 kcal was recorded.
Adherence to physical activity recommendations | Months 2, 4, and 6
  Physical activity and sedentary time will be measured objectively through a 7-day accelerometry protocol using ActiGraph wGT3X-BT (Pensacola, FL) accelerometers. Physical activity intensity will be scored based on established cutpoints, and minutes of moderate-vigorous physical activity (counted in bouts of ≥10 mins) will be calculated on each day of the assessment period.
Frequency of dietary lapses | Months 2, 4, and 6
  The occurrence of dietary lapses will be measured using ecological momentary assessment. Based on prior work, lapses are defined as "eating or drinking likely to cause weight gain, and/or put weight loss/maintenance at risk." If a lapse is endorsed at a given ambulatory assessment, subjects will classify them into one of four non-exclusive subtypes: (1) eating large portions, (2) eating at unplanned times, (3) eating foods inconsistent with weight control, or (4) eating when not hungry.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will develop an accessible archive of study data. After the study investigators have had a reasonable period of time to prepare manuscripts, study data sets will be stripped of all personal health information (PHI) to allow sharing of data without compromising subject confidentiality, privacy, and safety. All identification covered under HIPAA will be removed. A data sharing agreement will be required that will describe the conditions and restrictions of data use by external investigators; limited data access will be made available only to those users who successfully complete a rigorous approval process by the investigators.

DOCUMENTS (1):
  • Informed Consent Form (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT05326477/ICF_000.pdf